CLINICAL TRIAL: NCT04471350
Title: Post-market Evaluation of HEMOBLAST™ Bellows Performance and Safety in Spine Surgery
Brief Title: Post-market Evaluation of HEMOBLAST™ Bellows in Spine Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Indication withdrawn
Sponsor: Biom'Up France SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: ETC 2018-004
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Hemostasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: HEMOBLAST™ Bellows — Surgeon has chosen to use HEMOBLAST™ Bellows as an adjunct to hemostasis when control of minimal, mild, or moderate bleeding by conventional procedures is ineffective or impractical in spine surgery.

SUMMARY:
Prospective, multi-center, multi-national post-market study evaluating the performance and safety HEMOBLAST™ Bellows in spine surgery

DETAILED DESCRIPTION:
Prospective, multi-center, multi-national post-market study evaluating the performance and safety HEMOBLAST™ Bellows in spine surgery. Up to 80 subjects will be enrolled at up to 6 sites.

ELIGIBILITY:
Pre-operative Inclusion Criteria:

* Patient is undergoing a non-emergent spine surgery
* Patient is willing and able to give prior written informed consent for investigation participation;
* Patient is 18 years of age or older.

Intra-operative Inclusion Criteria

* Patient has one or more target bleeding sites (TBS) for which control of bleeding by conventional procedures is ineffective or impractical.
* The TBS(s) has been treated with HEMOBLAST™ Bellows per instructions for use.

Exclusion Criteria:

* Patient is pregnant, planning on becoming pregnant during the follow-up period, or actively breast-feeding;
* Patient has a known sensitivity or allergy to bovine and/or porcine substance(s) or any other component(s) of the hemostatic agent;
* Patient has religious or other objections to porcine, bovine, or human components;
* Patient has any other contraindications, warnings, precautions of the Approved Instruction For Use of HEMOBLAST™ Bellows preventing his/ her inclusion
* Patient is not appropriate for inclusion in the clinical trial, per the medical opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing spine surgery that meet all of the inclusion criteria and none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Achievement of Hemostasis | Intraoperatively, expected within 3-10 minutes of application
  The proportion of subjects for which hemostasis was achieved after application of HEMOBLAST™ Bellows.

SECONDARY OUTCOMES:
Incidence of Serious Adverse Device Effects (SADEs) | 4 weeks +/- 2 weeks
  The rate of occurrence of serious adverse events deemed by the Investigator to be possibly, probably, or definitely related to HEMOBLAST™ Bellows
Re-bleeding at Target Bleeding Site | Intraoperative, prior to surgical closure of the subject
  The rate of target bleeding site re-bleeding after hemostasis has been achieved with HEMOBLAST™ Bellows
Re-operation due to bleeding | Post-operatively, expected within 1-28 days of the surgical procedure
  The rate of re-operation due to post-operative bleeding/hemorrhage after treatment with HEMOBLAST™ Bellows

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie Longis, MD, Principal Investigator — L'Hôpital privé du Confluent
Locations (1):
- L'Hôpital privé du Confluent, Nantes, France

IPD SHARING:
Plan to Share IPD: No